CLINICAL TRIAL: NCT06891807
Title: RobAR Study: Comparison of Image Based Robotic TKA vs Imageless Augmented Reality-Assisted TKA
Brief Title: Comparison of Image Based Robotic Total Knee Arthroplasty vs Imageless Augmented Reality Assisted Total Knee Arthroplasty
Acronym: RobAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Centrum Latem (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Principal Investigator, Philippe Van Overschelde, Dr. Philippe Van Overschelde, MD, Orthopaedic Surgeon, Medisch Centrum Latem
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMS.2024.021; B0172024000001 (Other: AZMM)
Record Dates: First submitted 2024-12-05; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty(TKA); Total Knee Replacement Surgery
Keywords: Total Knee Arthroplasty (TKA); Knee Osteoarthritis; Assistive Technologies; Robotics; Augmented Reality
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Skywalker (Active Comparator): SkywalkerTM Robotics Assisted TKA using Evolution Medial Pivot Knee
  Interventions: Device: Robotics Assisted TKA
- Pixee Knee+ (Active Comparator): PIXEE Knee+ TKA using Evolution Medial Pivot Knee
  Interventions: Device: Augmented Reality assisted TKA

INTERVENTIONS:
Device: Robotics Assisted TKA — Skywalker Robotics Assisted TKA using Evolution Medial Pivot Knee
  Other Names: Skywalker Robotics Assisted TKA
  Arms: Skywalker
Device: Augmented Reality assisted TKA — Pixee Knee+ assisted TKA using Evolution Medial Pivot Knee
  Other Names: Pixee Knee+ TKA
  Arms: Pixee Knee+

SUMMARY:
This study compares the accuracy of two different techniques in placing a total knee replacement. In one technique, accurate instrument placement is facilitated by a robot, and in the other technique, augmented reality is used for correct instrument placement. Both surgical techniques are already commonly used. During both the robotic technique and the augmented reality technique, the additional information (angles - axes) obtained during the operation is used to optimize the placement of the various prosthesis components.

Patients that were recently diagnosed with advanced osteoarthritis of the knee can participate in this study. This means that the cartilage of the knee is affected by wear and tear. This causes pain, stiffness and swelling resulting in reduced mobility. When non-operative treatments are insufficient in treating the osteoarthritis, surgery is proposed wherein a knee arthroplasty is performed.

The goal of this study is to further optimize and personalize patient care. Additionally, the aim of the study is to investigate whether both techniques are equivalent in optimally placing the prosthesis and whether both techniques lead to comparable results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 18 years up to 85 years old
* Patients eligible and planned for a primary Total Knee Arthroplasty
* Patients willing to sign the informed consent form (ICF) for participating in this study
* Indication of surgery is primary osteoarthritis

Exclusion Criteria:

* Revision knee surgery
* Other medical conditions contributing to the rehabilitation process of the TKA according to the surgeon, such as Parkinson's Disease, dementia, multiple sclerosis and cerebral vascular accident
* The patient received a TKA within the last three months or has a TKA planned in the next three months, for the contralateral knee
* Patient is participating in another clinical trial
* Patient is not able to understand Dutch, French or English
* Patients who did not meet all of the inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
radiographic alignment and positioning of the implant on full-leg standing X-Rays | 1 year follow-up
  To evaluate the radiographic alignment and positioning of the implant on full-leg standing X-Rays at a minimum of 1 year follow up between two TKA assistive technologies. These results will be compared with the intraoperative settings for alignment and positioning of the implant.

SECONDARY OUTCOMES:
Safety and clinical outcomes of assistive TKA technologies | 2 year follow-up
  Percentage change from baseline in activity parameters measured by a wearable device and clinical status measured by patient reported outcome measurements (PROM) at 6 weeks, 3 months, 6 months, 1 year and 2 years after TKA surgery. Safety will be assessed based on the incidence of treatment-related complications (e.g., wound complications, infection, nerve injury, peri-prosthetic fracture, urinary tract infection, deep vein thrombosis and pulmonary embolism ) as reported by patients and documented in medical records.
Activity parameters | 2 year follow-up
  Percentage change from baseline in activity parameters (e.g., step count, activity types, amount of activities) measured by a wearable device, daily questionnaires and measured by the UCLA activity score at 6 weeks, 3 months, 6 months, 1 year and 2 years after TKA surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Medisch Centrum Latem, Sint-Martens-Latem, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No